CLINICAL TRIAL: NCT00567229
Title: Phase II Study of Lenalidomide and Rituximab for Patients With Relapsed and/or Refractory CD20+ Multiple Myeloma
Brief Title: Lenalidomide and Rituximab in Treating Patients With Recurrent and/or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mskcc 07-070; P30CA008748 (NIH); MSKCC-07070; NCT00590486 (obsolete NCT alias)
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Rituximab; Lenalidomide; Microarray Analysis; Flow Cytometry

ARMS (1):
- Lenalidomide and Rituximab (Experimental): This study will employ a Simon optimal two-stage design. Patients will receive lenalidomide 25 mg daily for days 1-21 of each 28 day cycle. Rituximab 375 mg/m2 will be given weekly for 4 weeks beginning 1 week after the start of lenalidomide therapy (weeks 2-5), and then once 8 weeks later (week 13). Patients with stable disease or better after 4 cycles (week 16, in the absence of delays for toxicity) will be able to continue on therapy on the same lenalidomide schedule and with rituximab 375 mg/m2 given once every 8 weeks.
  Interventions: Biological: rituximab; Drug: lenalidomide; Genetic: microarray analysis; Other: flow cytometry; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab
Drug: lenalidomide
Genetic: microarray analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving lenalidomide together with rituximab may be an effective treatment for multiple myeloma.

PURPOSE: This phase II trial is studying the side effects of giving lenalidomide together with rituximab and to see how well it works in treating patients with recurrent or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and efficacy, as determined by response rate (complete response [CR] + near CR + partial response), of lenalidomide administered with rituximab in patients with relapsed and/or refractory CD20+ multiple myeloma.

Secondary

* To assess the effects of this regimen on patient lymphocyte subsets (T, B, and NK cells) in peripheral blood and bone marrow samples from these patients.
* To perform detailed phenotypic analyses of NK cells in patient blood and bone marrow samples at baseline and post-treatment.

OUTLINE: Patients receive oral lenalidomide once daily on days 1-21. Treatment with lenalidomide repeats every 28 days for at least 4 courses. Patients also receive rituximab IV once weekly in weeks 2-5 and in week 13. Patients with stable disease then receive rituximab once every 8 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Peripheral blood samples are collected at baseline, and after courses 2 and 4. Samples are examined by flow cytometry for lymphocyte subset analysis (T-, B-, and NK-cell percentages and absolute numbers) and NK-cell phenotyping (CD16, CD56, NKG2D expression). Samples are also examined by immunologic assays of isolated peripheral blood mononuclear cells. Bone marrow aspirate samples are also collected at baseline and after course 2. Bone marrow mononuclear cells are isolated and evaluated by CD138+ plasma cell selection, ex vivo antibody-dependent cellular cytotoxicity assays, and bone marrow lymphocyte subset analysis.

After completion of study therapy, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD20+ multiple myeloma

  * CD20+ disease defined as co-expression of CD20 on ≥ 25% of the clonal plasma cell population as defined by immunohistochemical or flow cytometric staining of a bone marrow or plasmacytoma specimen obtained at study entry

    * For flow cytometry, this is determined by calculating the frequency of CD20+ CD138+ double-positive cells within the total CD138+ plasma cell population
    * For immunohistochemistry, this is determined by dual staining for CD20 and the involved clonal light chain (kappa or lambda), with a determination of the percent double-positive (≤ 25% or ≥ 25%)
* Symptomatic multiple myeloma that has relapsed or progressed after at least 1 prior anti-myeloma therapeutic regimen

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 16 weeks (4 months)
* ANC ≥ 1,500/μL (unless low ANC due to multiple myeloma)
* Platelets ≥ 100,000/μL (unless low platelets are due to multiple myeloma)
* Serum bilirubin ≤ 2.0 mg/dL
* AST, ALT, and alkaline phosphatase < 3 times upper limit of normal
* Serum creatinine ≤ 2.5 mg/dL
* Able to understand the investigational nature of lenalidomide and rituximab combination therapy and to give informed consent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception at least 28 days before, during, and for at least 28 days after completion or discontinuation of study treatment
* Able to take acetylsalicylic acid (ASA) (325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin)
* Prior malignancies with a disease free interval of ≥ 5 years allowed
* No history of thromboembolic disease within the past 6 months, regardless of anticoagulation
* No myocardial infarction within the past 6 months
* No New York Hospital Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No active hepatitis B or C infection
* No HIV 1or 2 positivity
* No acute ischemia or active conduction system abnormalities as evidenced by ECG
* No history of hypersensitivity reactions to lenalidomide, thalidomide, or rituximab
* No other medical condition or laboratory evaluation that, in the treating physician's or principal investigators' opinion, makes the patient unsuitable to participate in this clinical trial
* No concurrent active malignancy other than nonmelanoma skin cancers or carcinoma-in-situ of the cervix

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior therapy, including radiotherapy
* Prior lenalidomide or thalidomide allowed
* No prior rituximab

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hani Hassoun, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide and Rituximab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide and Rituximab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Final Response Rate After 4 Courses of Treatment
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Rituximab
Number analyzed (Participants) | 3
participants
  Stable Disease (SD) | 2
  Progression of Disease (POD) | 1

ADVERSE EVENTS:
Arm/Group | Lenalidomide and Rituximab
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Rituximab (N=3)
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Rituximab (N=3)
Constipation (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
PT INR (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes